CLINICAL TRIAL: NCT07338110
Title: Prospective Cohort Study of Patients Undergoing Surgical Repair of the Achilles Tendon
Brief Title: French Achilles Tendon Surgery Cohort Study
Acronym: AchilleCDS
Status: Recruiting | Type: Observational
Sponsor: Chirurgie Du Sport (Other)
Responsible Party: Principal Investigator, HARDY Alexandre, Surgeon, Chirurgie Du Sport
Other Study IDs: AchilleCDS
Record Dates: First submitted 2026-01-03; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Achilles Injuries Tendon; Surgery
Keywords: orthopedy; surgery; achille tendon repair; arthroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Achilles Tendon Surgery — Achilles tendon repair involves reattaching the torn ends of the tendon to restore its continuity and functional tension. This technique is typically used for acute ruptures where the tendon quality is preserved and direct suture is feasible.
  Achilles tendon reconstruction is performed in chronic ruptures, re-ruptures, or cases with significant tendon degeneration or retraction, where direct repair is not possible. The procedure may involve tendon transfers such as the flexor hallucis longus (FHL), or autografts from the triceps surae aponeurosis or hamstring tendons (gracilis-semitendinosus, DIDT). These techniques aim to restore tendon length, strength, and function.
  In some cases, augmentation techniques (e.g., pedicled or free grafts) are used to reinforce the repair, particularly in patients with poor tendon tissue quality or high functional demands.

SUMMARY:
This 20-year prospective cohort study monitors patients following Achilles tendon repair to assess re-rupture rates, long-term functional outcomes, return-to-sport rates, and procedure-related complications. The aim is to better understand the long-term durability and clinical effectiveness of Achilles tendon repair techniques to optimize patient outcomes.

DETAILED DESCRIPTION:
This study is a long-term cohort analysis involving patients who have undergone Achilles tendon repair surgery.

The goal is to follow these patients over a 20-year period to assess several key outcomes. Specifically, the study aims to evaluate the rate of re-ruptures, the rate and quality of return to sport, long-term functional outcomes using validated scoring systems, and the incidence of procedure-related complications.

By collecting detailed and consistent data over two decades, this research seeks to provide valuable insights into the durability and effectiveness of Achilles tendon repair surgery, ultimately contributing to a better understanding of the procedure and improved patient care.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing Achilles tendon repair surgery

Exclusion Criteria:

* Patient refusal

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients enrolled in the Achilles CDS cohort by one of the surgeons of the Chirurgie du Sport and meeting eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2043-04-01 (Estimated); Study Completion 2063-04-01 (Estimated)

PRIMARY OUTCOMES:
Re-rupture of the Achilles tendon | From the surgery to the end of the study (20years of follow-up for each patient)

SECONDARY OUTCOMES:
Return to sport | From the surgey to the end of follow up (20 years)
  Return to sport after surgery with the level of return, the type of sport and the delay. Questions regarding the return to sport at 6 months, 1 year, 2 years and every 2 years
Visual Analogue Scale | From the surgery to the and of the follow-up (20 years for each patient)
  The VAS score (Visual Analogue Scale) is a simple and widely used method for assessing subjective experiences, such as pain intensity, fatigue, or discomfort. It typically consists of a horizontal or vertical line, usually 10 cm in length, with endpoints representing the extremes of the experience being measured: 0: "No pain" (or "no discomfort"). 10: "Worst pain imaginable" (or "maximum discomfort") Evaluated during the 3 first days after surgery, at 6 months, 1 year, 2 years and every 2 years
Ankle Ligament Reconstruction - Return to Sport Injury score | From the surgery to the end of foolow-up (20 years for each patient)
  The ALR-RSI (Ankle Ligament Reconstruction - Return to Sport Injury) score is used to assess the patient's psychological state and apprehension regarding their return to sports activities. The score ranges from 0% (the lowest level of psychological readiness) to 100% (the highest level of psychological readiness). Questionnairy at 6 months, 1 year, 2 years and every 2 years
Foot an Ankle Ability Measure | From the surgery to the end of follow-up (20 years for each patient)
  Foot and Ankle Ability Measure (FAAM) is a tool designed to assess a patient's functional abilities and symptoms specifically related to their foot and ankle during daily activities and sports. It consists of two subscales: Activities of Daily Living (ADL): 21 items. Sports: 8 items. Each item is rated on a 5-point Likert scale: 4 = No difficulty 3 = Slight difficulty 2 = Moderate difficulty 1 = Extreme difficulty 0 = Unable to perform Scoring : Add the scores for all items within the subscale to calculate the total item score. Multiply the total number of answered items by 4 to determine the highest potential score (e.g., 84 for ADL and 32 for Sports if all items are answered). Divide the total item score by the highest potential score and multiply by 100. This gives the FAAM score, which ranges from 0% (lowest function) to 100% (highest function). Interpretation : A higher score indicates a greater level of physical function. Measured at 6 months, 1 year, 2 years and every 2 years
Achilles Tendon Total Rupture Score | From the surgery to the end of follow-up (20 years for each patient)
  The ATRS (Achilles Tendon Total Rupture Score) is used to assess the patient's functional recovery and ability to return to sports and daily activities after Achilles tendon rupture or surgery. The score ranges from 0 (severe limitations) to 100 (full recovery and no functional limitation). The questionnaire is administered at 6 months, 1 year, 2 years, and every 2 years thereafter.
UCLA Activity Scale | From the surgery to the end of follow-up (20 years for each patient)
  The UCLA Activity Score is used to assess the patient's general activity level and participation in sports or recreational activities after Achilles tendon injury or surgery. The score ranges from 1 (wholly inactive, dependent on others) to 10 (regular participation in impact sports). The questionnaire is administered at 6 months, 1 year, 2 years, and every 2 years thereafter.
Tegner Activity Scale | From the surgery to the end of follow-up (20 years for each patient)
  The Tegner Activity Scale is used to evaluate the patient's activity level, particularly in relation to sports and occupational demands, following Achilles tendon rupture or repair. The scale ranges from 0 (sick leave or disability due to knee/ankle injury) to 10 (competitive sports at elite level). The questionnaire is administered at 6 months, 1 year, 2 years, and every 2 years thereafter.
Post-Operative Joint Value | From the surgery to the end of follow-up (20 years for each patient)
  The Post-Operative Joint Value (PJV) is used to assess overall ankle function and patient satisfaction following Achilles tendon repair or reconstruction. The score combines objective measures (range of motion, stability) and patient-reported outcomes (pain, functional limitations). The scale typically ranges from 0 (poor joint function) to 100 (excellent joint function). The assessment is performed at 6 months, 1 year, 2 years, and every 2 years thereafter.
Complications | From the surgery to the end of follow-up (20 years for each patient)
  Complications after surgery recorded include, but are not limited to:
  * Removal of hardware
  * Infection
  * Hematoma
  * Re-repair of the Achilles tendon
  * Surgery for Achilles tendinopathy
  * Any other complications reported by the patient

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Hardy, MD, Principal Investigator — Chirurgie Du Sport
Locations (1):
- Chirurgie du Sport, Paris, Île-de-France Region, France